CLINICAL TRIAL: NCT02096107
Title: Safety and Efficacy of Everolimus Transition in Minimizing Progressive Graft Dysfunction and Interstitial Fibrosis in Adult Kidney Transplant Recipients
Brief Title: Novartis Everolimus Transition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00030099
Record Dates: First submitted 2014-02-28; First posted 2014-03-26 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Graft Dysfunction; Interstitial Fibrosis
Keywords: Everolimus; Graft dysfunction; Interstitial fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — Everolimus; Standard of Care

ARMS (2):
- Low intensity Tacrolimus (Active Comparator): Low tacrolimus, everolimus, and steroids
  Interventions: Drug: Everolimus
- Standard of Care (Other): Tacrolimus, mycophenolate mofetil and steroids
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Everolimus — Convert mycophenolate to everolimus with subsequent reduction in exposure to tacrolimus
  Arms: Low intensity Tacrolimus
Other: Standard of Care — Tacrolimus, mycophenolate mofetil and steroids
  Arms: Standard of Care

SUMMARY:
Transition from tacrolimus based triple therapy with Mycophenolate Mofetil (MMF) and steroids in stable renal transplant patients to low intensity tacrolimus, everolimus and prednisone will be associated with improvement in Glomular Filtration Rate (GFR) and allograft fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age and able to give informed consent.
2. Received a first or repeat cadaveric (including ECD) or living donor renal transplant.
3. Patient has stable graft function, defined as no change of greater than 40% of baseline serum creatinine and no acute rejection during the past month.
4. Currently receiving tacrolimus, mycophenolate mofetil and prednisone as their immunosuppression regimen

Exclusion Criteria:

1. Biopsy proven acute rejection episode that occurred within the past month.
2. Malignancy within the past 3 years, except for non-melanoma skin cancer.
3. Currently enrolled in an investigational drug trial.
4. Woman of child bearing potential not utilizing an effective form of birth control.
5. Patients with uncontrolled dyslipidemia, defined at serum fasting LDL >200 mg/dL or serum fasting triglycerides >500 mg/dL.
6. Patients with a spot urine protein to creatinine ratio of > 800 mg of protein per gram of creatinine.
7. WBC < 2,000 cells/mm3
8. Platelets < 75,000 cells/mm3
9. Patients who have received an organ transplant other than a kidney.
10. Patients with a history of biopsy proven FSGS, MPGN, or PGN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Titte Srinivas, MD, Principal Investigator — Medical University of South Carolina; David Taber, Principal Investigator — Medical University of South Carolina, Department of Surgery
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Taber DJ, Chokkalingam A, Su Z, Self S, Miller D, Srinivas T. Randomized controlled trial assessing the impact of everolimus and low-exposure tacrolimus on graft outcomes in kidney transplant recipients. Clin Transplant. 2019 Oct;33(10):e13679. doi: 10.1111/ctr.13679. Epub 2019 Sep 12. PMID 31365151

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Intensity Tacrolimus: Low tacrolimus, everolimus, and steroids
  Convert mycophenolate to everolimus (concentration goal of 3-8 ng/mL) with subsequent reduction in exposure to tacrolimus (concentration of 2-5 ng/mL)
- Standard of Care: Tacrolimus, mycophenolate mofetil and steroids
  Standard of Care: Tacrolimus (concentration goal of 5-12 ng/mL), mycophenolate mofetil and steroids
Period: Overall Study
Arm/Group | Low Intensity Tacrolimus | Standard of Care
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Intensity Tacrolimus | Standard of Care | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (13.6) | 51.6 (12.1) | 51.3 (12.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 11 | 14
  Male | 27 | 19 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 19 | 34
  White | 15 | 11 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 89.1 (17) | 84.7 (16.6) | 86.9 (16.8)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.6 (4.8) | 28.7 (4.5) | 28.7 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Kidney Allograft Fibrosis Assessment
Description: Measure and compare the change in interstitial fibrosis (morphometric analysis of trichrome stained slides) at one-year post-transplant in patients converted to everolimus, low intensity tacrolimus and prednisone versus the standard of care tacrolimus, mycophenolate and prednisone regimen.
  The scale is a percentage of the tissue that demonstrates fibrosis. The scale range is 0 to 100%. The higher the percentage, the worse the fibrosis and the poorer the prognosis. A lower score (percentage) is therefore better.
Time Frame: 1 year
Population: The number of subjects analyzed for the fibrosis assessment was 15 in each group, because biopsy samples for both baseline and end of follow-up were only able to be obtained from 15 subjects per group.
Measure: Mean (Inter-Quartile Range); unit: % of fibrosis
Arm/Group | Low Intensity Tacrolimus | Standard of Care
Number analyzed (Participants) | 15 | 15
% of fibrosis
  Baseline | 22.9 [17.9 to 25.7] | 20.8 [18.4 to 30.4]
  End of Follow-up | 22.9 [18.6 to 28.1] | 27.8 [18.7 to 31.0]

2. Secondary Outcome: Renal Function Measured by Estimated Glomerular Filtration Rate (eGFR)
Description: Measure and compare the estimated GFR (using the 4-variable modified MDRD equation) in patients converted to everolimus, low intensity tacrolimus and prednisone versus the standard of care tacrolimus, mycophenolate and prednisone regimen, both at one year and two years post-transplant.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Low Intensity Tacrolimus | Standard of Care
Number analyzed (Participants) | 30 | 30
mL/min/1.73 m^2 | 59 (14) | 56 (15)

3. Secondary Outcome: Kidney Allograft Survival
Description: Compare the patient and graft survival rates at one-year post-transplant in each group.
Time Frame: 1 year
Measure: Number; unit: percentage of patients graft survival
Arm/Group | Low Intensity Tacrolimus | Standard of Care
Number analyzed (Participants) | 30 | 30
percentage of patients graft survival | 100 | 100

4. Secondary Outcome: Percentage of Participants Discontinuing or Modifying Immunosuppressant Use
Description: Measure and compare the rates of immunosuppressant discontinuation and modification for each group.
Time Frame: 2 year
Measure: Number; unit: percentage of participants
Arm/Group | Low Intensity Tacrolimus | Standard of Care
Number analyzed (Participants) | 30 | 30
percentage of participants | 37 | 20

5. Secondary Outcome: Adverse Drug Reactions
Description: Measure and compare the incidence of significant immunosuppressant-related adverse drug reactions for each group.
Time Frame: 2 year
Measure: Count of Participants; unit: Participants
Arm/Group | Low Intensity Tacrolimus | Standard of Care
Number analyzed (Participants) | 30 | 30
Participants | 11 | 6

6. Secondary Outcome: Infection
Description: Compare the rates of post-transplant infections, including CMV, BK, and admissions to the hospital for infectious causes in each group.
Time Frame: 2 year
Measure: Number; unit: percentage of subjects with infection
Arm/Group | Low Intensity Tacrolimus | Standard of Care
Number analyzed (Participants) | 30 | 30
percentage of subjects with infection | 17 | 30

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Low Intensity Tacrolimus | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 8/30 | 6/30
Other Adverse Events (participants affected / at risk) | 11/30 | 6/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Intensity Tacrolimus (N=30) | Standard of Care (N=30)
Hospitalization (Renal and urinary disorders) | 8 (8) | 6 (6) — Post-randomization hospitalization occurrence
Infections (Renal and urinary disorders) | 4 (4) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Intensity Tacrolimus (N=30) | Standard of Care (N=30)
Immunosuppression held or modified (Renal and urinary disorders) | 11 (11) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-30): https://cdn.clinicaltrials.gov/large-docs/07/NCT02096107/Prot_SAP_000.pdf